CLINICAL TRIAL: NCT02399644
Title: Physical Activity and Acceptance and Commitment Therapy as Treatment for Long Term Pain. A Randomized Controlled Trial
Brief Title: Physical Activity and Acceptance and Commitment Therapy as Treatment for Long Term Pain
Acronym: FACTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Bjorn Gerdle, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REHSAM_RS2010/002
Record Dates: First submitted 2015-01-21; First posted 2015-03-26 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2015-03

CONDITIONS: Chronic Pain
Keywords: pain; rehabilitation; exercise; psychological; intervention
MeSH Terms: conditions — Chronic Pain; Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ACT (Experimental): Acceptance and Commitment Therapy is a version of Cognitive behavioral Therapy that focuses on acceptance and mindfulness. The aim is to prevent avoidance and control of negative private events such as anxiety or pain. The treatment consists of 7 weekly group sessions, 2 hours a week. The participants are given homework between sessions.
  Interventions: Behavioral: ACT
- Physical activity (Experimental): Participants are going to participate in a training programme including aerobic exercise as well as endurance and strength training for the neck, shoulders, low back, core and leg muscles. The training is group-based and supervised by a physiotherapist two times a week, one hour a time for eight weeks. Home exercises twice a week are also a part of the intervention. It is possible to individually adjust movements and intensity to the participants' capacity if needed.
  Interventions: Other: Physical activity
- Experience based discussion group (No Intervention): Participants are going to discuss their experiences of long term pain. The discussions is supervised by a heath care professional and is based on beforehand defined subjects, i.e. relations, spare time, economics, occupation. The meetings are hold for 7 weeks, 2 hours a week.

INTERVENTIONS:
Behavioral: ACT — ACT is a type of Cognitive behavioral Therapy (CBT) that focuses on acceptance and mindfulness. The aim is to prevent avoidance and control of negative private events such as anxiety or pain. The treatment consists of 7 weekly group sessions, 2 hours a week. The participants are given homework between sessions.
  Arms: ACT
Other: Physical activity — Participants are going to perform a training programme including aerobic exercise as well as endurance and strength training for the neck, shoulders, low back, core and leg muscles. The training is group-based and supervised by a physiotherapist two times a week, one hour a time for eight weeks. Home exercises twice a week are also a part of the intervention. It is possible to individually adjust movements and intensity to the participants' capacity if needed.
  Arms: Physical activity

SUMMARY:
Only to a limited extent has been compared the effectiveness of physical exercise and psychological interventions in subjects with chronic pain. Knowledge about this is necessary in order to compose optimal multimodal rehabilitation programs at different health care levels. Moreover, assuming that both types of interventions have effects, these effects may necessarily not concern the same outcome variables. Therefore it may be important to understand to what extent the effects overlap and the extent to which the effects are isolated to an intervention.

The overall strategic purpose of the present study is to develop effective multimodal rehabilitation programs. In this study the effectiveness of following three interventions are compared.

* Group-based rehabilitation according to a concept based on an Acceptance and Commitment Training -Stress Management Intervention (ACT-SMI)
* Group-based rehabilitation compromised of physical exercise (Exercise).
* Group-based discussion concerning pain and its consequences (i.e., the control group, CON) The effectiveness is investigated with respect to long-term effects on pain and its consequences, including perceived health and return to work / sick leave.

The overall hypothesis is that the former intervention means better long-term results because it clearly helps the individual to process the psychological aspects of itself likely to have long lasting effects.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain in the neck and/or back with or without pain in one or more quadrants of the body

Exclusion Criteria:

* Inflammatory and neurological diseases, severe social and/or psychological problems, patients that already have taken part in multidisciplinary rehabilitation programs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity | Change from baseline pain intensity at 12 months
  Pain intensity recent 7 days using a numeric rating scale
Change in Depression | Change from baseline depression at 12 months
  Depression scale of Hospital Anxiety and Depression Scale (HADS)
Change in Catastrophizing | Change from baseline catastrophizing at 12 months
  The Pain Catastrophizing Scale (PCS)
Change in Acceptance | Change from baseline acceptance at 12 months
  The Chronic Pain Acceptance Questionnaire (CPAQ)
Change in Disability | Change from baseline disability at 12 months
  Pain Disability Index (PDI)

SECONDARY OUTCOMES:
Change in Flexibility | Change from baseline flexibility at 12 months
  The Psychological Inflexibility in Pain Scale (PIPS)
Change in Insomnia | Change from baseline insomnia at 12 months
  The Insomnia Severity Index (ISI)
Change in Fear-avoidance beliefs | Change from baseline fear-avoidance at 12 months
  Fear-Avoidance Beliefs Questionnaire (FABQ)
Change in Disability2 | Change from baseline disability2 at 12 months
  Oswestry Disability Index (ODI)
Change in Health | Change from baseline health at 12 months
  The EuroQol instrument
Change in Life satisfaction | Change from baseline life satisfaction at 12 months
  The Life Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Gerdle, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Rehabilitation medicine, IMH, Linköping University, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Wiklund T, Linton SJ, Alfoldi P, Gerdle B. Is sleep disturbance in patients with chronic pain affected by physical exercise or ACT-based stress management? - A randomized controlled study. BMC Musculoskelet Disord. 2018 Apr 10;19(1):111. doi: 10.1186/s12891-018-2020-z. PMID 29631567